CLINICAL TRIAL: NCT00325780
Title: Open-Label, Long-Term (1 Year) Extension Study of Pitavastatin in Patients With Primary Hypercholesterolemia or Combined Dyslipidemia
Brief Title: Long-Term Extension Study of Pitavastatin in Patients With Primary Hypercholesterolemia or Combined Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Research Europe (Industry)
Responsible Party: Dragos Budinski, MD, Kowa Research Europe
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK-104-307; 2005-001112-41
Record Dates: First submitted 2006-02-10; First posted 2006-05-15 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Hypercholesterolemia; Dyslipidemia
Keywords: Kowa; Hypercholesterolemia; dyslipidemia; pitavastatin; NK-104; Hypercholesterolemia or combined dyslipidemia
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias | interventions — pitavastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pitavastatin 4 mg QD (Experimental): Pitavastatin 4 mg once daily
  Interventions: Drug: Pitavastatin

INTERVENTIONS:
Drug: Pitavastatin — Pitavastatin 4 mg once daily

SUMMARY:
This study is a long-term follow-up protocol for patients who participated in study NK-104-3.01EU or study NK-104-3.02EU.

DETAILED DESCRIPTION:
Patients from the NK-104-3.01EU and NK-104-3.02EU studies will continue to receive either pitavastatin or the comparator statin for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients have completed 12 weeks of treatment in Study NK-104-301 (NCT00249249) or NK-104-302 (NCT00309777)
* Patients who have not developed any treatment emergent and, in the opinion of the investigator, related adverse event (AE) of clinical significance where the investigator is uncomfortable with continuing the patient on therapy with pitavastatin.
* Patients who have been following a fat and cholesterol restrictive diet.

Exclusion Criteria:

* Any conditions which may cause secondary dyslipidemia should be reassessed at the beginning of the follow-up study.
* Uncontrolled diabetes mellitus should be reassessed at the beginning of the follow-up study.
* Abnormal pancreatic, liver, or renal function
* Abnormal serum ALAT/SGPT/ALT, ASAT/SGOT/AST, or creatine kinase (CK) above the pre-specified level
* Significant heart disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1355 (Actual)
Dates: Start 2006-07; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dragos Budinski, Med Dr., Study Director — Medical Director
Locations (186):
- Denmark (6):
  - Copenhagen University Hospital, Copenhagen
  - Medical Center, Copenhagen
  - Y Forskning, Bispebjerg Hospital, Copenhagen Nv
  - Frederiks Hospital, Kardiologisk, Frederiksberg
  - Kolesterollaboratoriet, Hellerup
  - CCBR A/S, Vejle
- Finland (5):
  - Geri-Med Oy, Helsinki
  - Kaisaniemen Laakariasema, Helsinki
  - Keravan Laakarikeskus, Helsinki
  - SOK-Tyoterveyshuolto, Tampere
  - TYKS University Hospital, Turku
- Germany (20):
  - Kardiologische Gemeinschaftspraxis Prof. Reifart, Bad Soden/Taunus
  - Praxis Dr. Boenninghoff, Beckum
  - Klinische Forschung Berlin Mitte, Berlin
  - Gemeinschaftspraxis am Bahnhof, Berlin-Spandau
  - Pharmakologisches Studienzentum Chemnitz, Chemnitz
  - GWT-TUK mbH, Zentrum fur Klinische Studien, Dresden
  - Internistische Diabetische Schwerpunktpraxis Dr., Frankfurt am Main
  - Gemeinschaftspraxis Dr. Krause, Th. Menke, Goch
  - Klinische Forschung Hamburg, Hamburg
  - Innere Medizin I/Medizinische Klinik, Heidelberg
  - Gemeinschaftspraxis H. Holz Dr. Med, K. W. Klingl, Lampertheim
  - ZET-Studien GmbH Leipzig, Leipzig
  - Internistische Gemeinschaftspraxis, Mainz
  - Praxis Dr. Wachter, Mannheim
  - Gemeinschaftspraxis Melcherstaette, Melcherstaette
  - Gemeinschaftspraxis Dr. Senftleber, Dr. Kohler, Messkirch
  - Praxisgemeinschaft im Kleinen Biergrund, Offenbach/M
  - Gemeinschaftspraxis Drs. Mockesch, Weinheim
  - Intermed Institud fur Klinische Forschung und Arzn, Wiesbaden
  - Gemeinschaftspraxis Dr. Emden, Frank Drewes, Worpswede
- India (18):
  - Care Hospital, Andhra Pradesh
  - School of Diabetology, Nizam Institute of Medical Sciences, Andhra Pradesh
  - Bhagwan Mahaveer Jain Heart Centre, Bangalore
  - Sri Ramachandra Medical College Hospital, Chennai
  - Heart Care Clinic, Gujarat
  - Apollo Hospitals, Hyderabad
  - CARE Group of Hospitals, Hyderabad
  - St. John's Medical College Hospital, Karnataka
  - Bathia Hospital, Maharashtra
  - LTMMC & General Hospital, Maharashtra
  - Sir J. J. Group of Hospitals, Maharashtra
  - King Edward Medical College & Hospital, Maharashtra
  - Ruby Hall Clinic, Maharashtra
  - Lokmanya Hospital, Maharashtra
  - PD Hinduja Hospital, Mumbai
  - Sir Gagaram Hospital, New Delhi
  - Apollo Hospital, Tamil Nadu
  - Department of Cardiology, Tamil Nadu
- Israel (9):
  - Department of Internal Medicine, Soroka Medical Center, Beersheva
  - Department of Internal Medicine A, Rambal Medical Center, Haifa
  - Department of Internal Medicine, Wolfson Medical Center, Holon
  - Center for Research, Hadassah University Hospital, Jerusalem Ein Kerem
  - Meir Hospital, Kfar Saba
  - Department of Medicine, Hadassah Medical Center, Mount Scopus Jerusalem
  - Department of Internal Medicine, Rivka Sieff Medical Center, Safed
  - Institute of Metabolic Diseases, Tel Aviv
  - Institute of Lipid & Atherosclerosis Research, Tel Litwinsky
- Italy (10):
  - Dipartimento di Medicina Clinica e Biotecnologia Applicata, Bologna
  - Centro di Ricerca Clinica, Chieti
  - Gerontologia e Geriatria - Universita degli Studi, Ferrara
  - Dipartimento di Medicina Interna DIMI, Genova
  - Universita di Modena e Reggio Emilia, Policlinico, Modena
  - Dipartimento di Medicina Clinica e Sperimentale, Napoli
  - Medicina Clinica e delle Patologie Emergenti, Palermo
  - Dipartimento di Medicina Interna e Scienze Biomediche, Parma
  - U.O. Malattie Metaboliche e Diabetologia, Treviglio
  - Azienda Ospedaliero-Universitaria, Trieste
- Netherlands (19):
  - Andromed Breda, Breda
  - Middellaan 5, Breda
  - Andromed Eindhoven, Eindhoven
  - Bomanshof 8, Eindhoven
  - Andromed Noord, Groningen
  - Damsterdiep 9, Groningen
  - Vasculair Onderzoek Centrum Hoorn, Hoorn
  - Andromed Leiden, Leiden
  - Doezastraat 1, Leiden
  - Andromed Nijmegen, Nijmegen
  - Kamerlingh Onnesstraat 16-18, Nijmegen
  - Andromed Rotterdam, Rotterdam
  - Mathenesserlaan 247, Rotterdam
  - Albert Schweitzer Ziekenhuis, Sliedrecht
  - Andromed Oost, Velp
  - Reigerstraat 30, Velp
  - Rivierenland Tiel, Wp Tiel
  - Andromed Zoetermeer, Zoetermeer
  - Parkdreef 142, Zoetermeer
- Norway (4):
  - Nyomen Legekontor, Kongsberg
  - Radhuset Spesialistsenter, Oslo
  - Rikshospitalet - University Hospital, Oslo
  - Skedsmo Medisinske Senter A.S., Skedsmokorset
- Poland (10):
  - Podlaski Osrodek Kardiologii, Bialystok
  - NZOZ GCP Dobra Praktyka Lekaska, Gruziadz
  - NZOZ Terapia Optima, Katowice
  - NZOZ Centrum, Poradnia Kardiologiczna, Siedlce
  - Spec. Gab. Lek. Internistyczno-Kardiologicznly, Tarnów
  - Woj.Szp.Spec.Nr 1 im. Prof. J. Gasinskiego, Tychy
  - Instytut Zywnosci i Zywienia, Warsaw
  - Lecznica PROSEN SMO, Warsaw
  - Szpital Wolski,im. Dr A. Gostynskiej, Warsaw
  - NZOZ Esculap, Przychodnia Lekary Rodzinnych, Łosice
- Russia (26):
  - Kemerovo Cardiology Dispensary, Kemerovo
  - Central Clinical Hospital 1 of RZD, Moscow
  - City Clinical Hospital 23, Moscow
  - City Clinical Hospital 64, Moscow
  - Federal State Institution Out-Patient Clinic ï€£3 of Russian Federation of Presidentâ€™s Management, Moscow
  - Moscow City Clinical Hospital 68, Moscow
  - Moscow Regional Research Clinic Institute n.a.M.F.Vladimirov, Department of Therapy, Moscow
  - State Educational Institution of Higher Professional Education â€œMoscow State University of Medicine and Dentistry of Federal Agency of Health Care and Social Developmentâ€�, Department of Internal Diseases and Rheumatology based at City Clinica, Moscow
  - State Educational Institution of Higher Professional Education â€œMoscow State University of Medicine and Dentistry of Federal Agency of Health Care and Social Developmentâ€�, Hospital Therapy Department # 1 based at City Clinical Hospital # 40, Moscow
  - State Educational Institution of Higher Professional Education â€œMoscow State University of Medicine and Dentistry of Federal Agency of Health Care and Social Developmentâ€�, Hospital Therapy Department #1 based at City Clinical Hospital # 52, Moscow
  - State Educational Institution of Higher Professional Education â€œRussian State Medical University Federal Agency of Health Care and Social Developmentâ€�, Department of Polyclinic Therapy based at Diagnostic Center # 1, Moscow
  - State Educational Institution of Higher Professional Education â€œRussian State Medical University Federal Agency of Health Care and Social Developmentâ€�, Department of Therapy based at City Hospital # 4, Moscow
  - State Educational Institution of Higher Professional Education â€œRussian State Medical University of Federal Agency of Health Care and Social Developmentâ€�, Department of Hospital Therapy #1 based at City Clinical Hospital #15, Cardiology Depar, Moscow
  - State Institution â€œResearch Institute of Physical and Chemical Medicineâ€� of Federal Agency of Health Care and Social Development, Laboratory of Clinical Cardiology based at Bauman City Hospital # 29, Moscow
  - State Institution â€œRussian Cardiology Research Complexâ€� of Federal Agency of Health Care and Social Development, Myasnikov Clinical Cardiology Institute, Department of Hemodialysis and Plasmapheresis, Moscow
  - State Research Center for Preventive Medicine, Moscow
  - Novosibirsk Reg. Clinical Cardiology Dispensary, Novosibirsk
  - Central Medical Unit 122, St. Pb, Saint Petersburg
  - Clinical Hospital of Russian Academy of Sciences, Saint Petersburg
  - Consulting and Diagnostic Center 85, Saint Petersburg
  - Krestovsky Island Medical Institute, Saint Petersburg
  - Pokrovskaya City Hospital, Saint Petersburg
  - St. Petersburg State Medical Institution â€œOut-patient Clinic # 109â€�, Saint Petersburg
  - St.Petersburg State Medical Institution â€œPokrovskaya City Hospitalâ€�, Cardiology Department #2, Saint Petersburg
  - State Educational Institution of Higher Professional Education, â€œSaint-Petersburg State Medical University n.a.Academician I.P.Pavlov of Federal Agency of Health Care and Social Developmentâ€�, Chair and Department of Faculty Therapy, Saint Petersburg
  - State Educational Institution of Higher Professional Education, â€œSaint-Petersburg State Medical University n.a.Academician I.P.Pavlov of Federal Agency of Health Care and Social Developmentâ€�, Institute of Cardiovascular Diseases, Saint Petersburg
- Spain (19):
  - Hospital Clinico S. Juan de Alicante, San Juan, Alicante
  - Hospital Clinic i Provincial, Villaroel, Barcelona
  - Hospital de San Vicente, Alicante
  - Hospital Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Ramon y Cajal, Madrid
  - Centro de Especialidades Pedro Gonzalez Bueno, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Centro de Salud de Ventanielles, Oviedo
  - Hospital Marques de Valdecilla, Santander
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital Virgen del Roci-o, Seville
  - Hospital Dr. Peset, Valencia
  - Hospital de Sagunto, Valencia
  - Hospital Clinico Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza
- Sweden (10):
  - Angelholms Sjukhus, Medicinkliniken, Angelhom
  - Sahlgrenska University Hospital, Intermedicin, Gothenburg
  - Hjartmottagningen, Helsingborg
  - Lakarcentrum Nyponet, Karineholm
  - Medicinkliniken, Ludvika
  - Huslakaren i Sandviken, Sandviken
  - Narsjukhuset Sandviken, Kardiologlab, Medicin, Sandviken
  - Hjart & Karlcenter, Södertälje
  - Karolinska Universitetssjukhuset, Stockholm
  - Hjarthuset AB, Varberg
- United Kingdom (30):
  - Oldfield Surgery, Bath
  - St James's Surgery, Bath
  - St Michael's Partnership, Bath
  - The Pulteney Practice, Bath
  - Birmingham Clinical Research Centre, Birmingham
  - Stonehill Medical Center, Bolton
  - Avondale Surgery, Chesterfield
  - Chorley Clinical Research Centre, Chorley
  - Saltash Health Center, Cornwall
  - Gomersal Lane Surgery, Dronfield
  - Townhead Research, Irvine
  - Crosby Clinical Research Centre, Liverpool
  - The Symons Medical Center, Maidenhead
  - Manchester Clinical Research Centre, Manchester
  - Greenwood Medical Center, Nottingham
  - Knowle House Surgery, Plymouth
  - Reading Clinical Research Centre, Reading
  - Elm Lane Surgery, Sheffield
  - The Burngreave Surgery, Sheffield
  - Brook Lane Surgery, Southampton
  - St Helier Hospital, Surrey
  - Box Surgery, Wiltshire
  - Bradford Road Medical Center, Wiltshire
  - Eastleigh Surgery, Wiltshire
  - Lovemead Group Practice, Wiltshire
  - Rowden Medical Partnership, Wiltshire
  - St Chad's Surgery, Wiltshire
  - The Health Centre, Wiltshire
  - The Porch Surgery, Wiltshire
  - The Burns Medical Practice, Yorkshire

REFERENCES:
- [Derived] Ose L, Budinski D, Hounslow N, Arneson V. Long-term treatment with pitavastatin is effective and well tolerated by patients with primary hypercholesterolemia or combined dyslipidemia. Atherosclerosis. 2010 May;210(1):202-8. doi: 10.1016/j.atherosclerosis.2009.12.009. Epub 2009 Dec 11. PMID 20080236

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pitavastatin 4 mg QD
Started | 1355
Safety Population | 1353 (Patients who received at least one dose of study treatment in this extension study.)
Completed | 1200
Not Completed | 155

BASELINE CHARACTERISTICS:
Arm/Group | Pitavastatin 4 mg QD
Number analyzed (Participants) | 1353
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 941
  >=65 years | 412
Age Continuous [Mean (Standard Deviation); unit: years] | 58.6 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 778
  Male | 575

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C)
Description: Mean percent change from baseline in low-density lipoprotein cholesterol (LDL-C)
Time Frame: Baseline to 52 Weeks
Population: Patients who had an observation at Week 52
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pitavastatin 4 mg QD
Number analyzed (Participants) | 1202
percent change | -42.89 (16.001)

2. Secondary Outcome: Change From Baseline in Total Cholesterol
Description: Mean percent change from baseline in total cholesterol
Time Frame: Baseline to 52 weeks
Population: Patients who had an observation at Week 52
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pitavastatin 4 mg QD
Number analyzed (Participants) | 1203
percent change | -29.59 (12.549)

ADVERSE EVENTS:
Arm/Group | Pitavastatin 4 mg QD
Serious Adverse Events (participants affected / at risk) | 49/1353
Other Adverse Events (participants affected / at risk) | 293/1353
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pitavastatin 4 mg QD (N=1353)
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 4
Atrial fibrillation (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 4
Ventricular extrasystoles (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Retinal detachment (Eye disorders) | 1
Diverticulum (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 1
Gastric polyps (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Cardiac death (General disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Anal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Chronic tonsillitis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Osteomyelitis acute (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Fascitis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cranial neuropathy (Nervous system disorders) | 1
Hypoxic encephalopathy (Nervous system disorders) | 1
Ischaemic cerebral infarction (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 2
Vascular encephalopathy (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1
Hypertension (Vascular disorders) | 2
Thrombophlebitis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pitavastatin 4 mg QD (N=1353)
Influenza (Infections and infestations) | 41
Nasopharyngitis (Infections and infestations) | 73
Arthralgia (Musculoskeletal and connective tissue disorders) | 46
Myalgia (Musculoskeletal and connective tissue disorders) | 55
Blood creatine phosphokinase increased (Investigations) | 78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days